CLINICAL TRIAL: NCT03672721
Title: A Phase II Study in Relapsing Glioblastoma of Intraarterial Concurrent Chemoradiation Therapy Using IA Carboplatin
Brief Title: IA Carboplatin + Radiotherapy in Relapsing GBM
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, David Fortin, full professor in surgery, Université de Sherbrooke
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2018-2452
Record Dates: First submitted 2018-07-11; First posted 2018-09-14 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma Multiforme; Relapse
MeSH Terms: conditions — Glioblastoma; Recurrence

STUDY DESIGN:
Intervention Model Description: Dose escalation study of combined intraarterial carboplatin + radiotherapy. Total number of 6 arms, 5 patients per arms plus 5 patients in the arm determined as the NOAEL: arm 1 = 400 mg/m^2 carbo + 15 Gy; arm 2 = 400 mg/m^2 carbo + 18 Gy; arm 3 = 400 mg/m^2 carbo + 20 Gy; arm 4 = 400 mg/m^2 carbo + 25 Gy; arm 5 = 400 mg/m^2 carbo + 30 Gy and arm 6 = 400 mg/m^2 carbo + 35 Gy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Arm 1: IA Carbo + radiation (Experimental): 400 mg/m^2 carbo + 15 Gy
  Interventions: Drug: IA Carbo+ Radiation
- Arm 2: IA Carbo + radiation (Experimental): 400 mg/m^2 carbo + 18 Gy
  Interventions: Drug: IA Carbo+ Radiation
- Arm 3: IA Carbo + radiation (Experimental): 400 mg/m^2 carbo + 20 Gy
  Interventions: Drug: IA Carbo+ Radiation
- Arm 4: IA Carbo + radiation (Experimental): 400 mg/m^2 carbo + 25 Gy
  Interventions: Drug: IA Carbo+ Radiation
- Arm 5: IA Carbo + radiation (Experimental): 400 mg/m^2 carbo + 30 Gy
  Interventions: Drug: IA Carbo+ Radiation
- Arm 6: IA Carbo + radiation (Experimental): 400 mg/m^2 carbo + 35 Gy
  Interventions: Drug: IA Carbo+ Radiation

INTERVENTIONS:
Drug: IA Carbo+ Radiation — combination of intraarterial carboplatin + radiation in dose escalation

SUMMARY:
Treatment of glioblastoma involves an optimal surgery, followed by a combination of radiation and temozolomide chemotherapy. Progression-free survival (PFS) with this treatment is only 6.9 months and relapse is the norm. The rationale behind the fact that limited chemotherapy agents are available in the treatment of malignant gliomas is related to the blood-brain barrier (BBB), which limits drug entry to the brain. Intraarterial (IA) chemotherapy allows to circumvent this. Using IA delivery of carboplatin, the investigators have observed responses in 70% of patients for a median PFS of 5 months. Median survival from study entry was 11 months, whereas the overall survival 23 months. How can this be improved? By coupling radiation with a chemotherapeutic which is also a potent radiosensitizer such as carboplatin.

Study design: In this phase I/II trial, patients will be treated at recurrence; a surgery will be performed for cytoreduction and to obtain tumor sample, followed with a combination of re-irradiation and IA carboplatin chemotherapy. A careful escalation scheme from 1.5Gy/fraction up to 3.5Gy/fraction will allow the investigators to determine the optimal re-irradiation dose (10 fractions of radiation over 2 weeks). Toxicity will be assessed according to the NCIC common toxicity criteria. Combined with radiation, patients will receive 2 treatments of IA carboplatin, 400 mg/m2, 4 hours prior to the first and the sixth radiation fraction. IA treatments will then be continued on a monthly basis, up to a total of 12 months, or until progression.

Outcome measurements: Tumor response will be evaluated using the RANO criteria by magnetic resonance imaging monthly. The investigators will also acquire a sequence that enables the measurement of cerebral blood flow, cerebral blood volume and blood vessel permeability that are all relevant to understand the delivery of therapeutics to the CNS. Primary outcome will be OS and PFS. Secondary outcome will be QOL, neurocognition, and carboplatin delivery.

In vitro intracellular carboplatin accumulation: Tumor samples from re-operation will be be analyzed for intracellular Pt concentration by ICP-MS. The amount of Pt bound to DNA will be measured. The level of apoptosis will be determined for each of the sample.

Putting together these data will allow to correlate clinical and radiological response to QOL, NC (MOCA), and to delivery surrogates for the IA infusion and intracellular penetration of carboplatin.

DETAILED DESCRIPTION:
A phase II study in relapsing glioblastomas (GBM) using concurrent intraarterial carboplatin chemoradiation therapy.

BACKGROUND - Contemporary treatment of GBM brain tumors involves a first-line treatment in which the patient receives a surgical procedure followed by a combination of radiation and temozolomide-based chemotherapy1. Unfortunately, this regimen improves patient survival only modestly, with a progression-free survival (PFS) of 6 months, and an overall survival of 14 months. Glioblastoma remains an incurable disease characterized by relapse and disease progression. There is no established second-line treatment for relapsing GBM, and the most used (BCNU chemotherapy) results in a PFS of only 2 months. As the investigators have shown, treatment can be considerably improved by circumventing the limitation of chemotherapeutic agents(CA) to cross the blood-brain barrier (BBB) and enter the central nervous system (CNS).

The investigators have focused their research on 3 essential aspects of GBM treatment: 1) alternate delivery approaches to bypass the BBB; 2) magnetic resonance imaging (MRI) to characterize tumor blood supply and predict therapeutics delivery to the tumor; 3) synergestic interplay of radiation and platinum drugs to improve brain tumor therapy. This is the first study to ever attempt bridging these 3 aspects within the same project.

Alternate delivery approaches to bypass the BBB.

Although different approaches have been tested in the researcher's lab to bypass the BBB, the most applicable to the clinic is the intraarterial infusion of chemotherapy (IA). It allows to circumvent the BBB via the first pass effect, resulting in a local plasma peak concentration increase of the CA by up to a 5-fold factor, maximizing CNS drug exposure. It also decreases systemic distribution of the CA thereby reducing toxicities and side effects. Over the last 15 years, the principal investigator has treated more than 720 patients using this IA approach, 422 of which had glioblastoma. This is the largest of such series. Based on this extensive experience, the investigators have convincingly shown that the procedure is safe and well tolerated. Using IA carboplatin in GBM relapse, a response in 70% of patients, and a 22 months overall survival + an increase in PFS to 5 months has been observed. This represents an impressive survival increase of 9 months. Time is ripe to improve these results in hope to cure this hard-to-treat cancer someday; hence the 2 additional measures discussed next.

MRI characterization. MRI is routinely used to monitor GBM response to treatment. This imaging procedure could also help guide treatment and predict responses. Indeed, the investigators have recently developed a novel MRI sequence that enables the simultaneous measurement of cerebral blood flow (CBF), cerebral blood volume (CBV) and vessel permeability; these surrogates are all relevant to predict delivery of therapeutics to CNS tumors. This sequence has been tested and has met strict quality criteria. This will help decide the artery into which IA chemotherapy is delivered, and predict CA delivery and possibly tumor response.

Synergistic interplay of radiation and platinum drugs. Radiotherapy is the most effective single-treatment modality for GBM tumors, but controls the disease only transiently. A way to improve treatment consists of coupling radiation with a potent radiosensitizer. Carboplatin (Ca), a platinum (Pt) drug, is ideally suited for this7. Our group has demonstrated that the addition of Ca to ionizing radiation produced significantly more DNA strand breaks. In numerous cell lines, combining radiotherapy and Ca was found to increase cell death. In a mouse model, the investigators observed a maximum antitumor effect with Pt-Ca administration at 4 h or 48 h prior to irradiation. This timing correlated to the highest levels of Pt bound to DNA. Concurrent Pt-Ca and radiation treatment represents a common modality for treating a variety of cancers. Unfortunately, since this class of drug does not readily cross the BBB when administered via the standard iv routes, such compounds are not used to treat GBM.

After years of interdisciplinary collaboration, the investigators demonstrated the following key factors in our pre-clinical F98-Fischer GBM model: 1- the use of the IA route increased Ca accumulation into the nucleus of tumor cells by a whooping 20-fold factor compared to the iv route. 2- While testing for 5 different Platinum compounds administered to the CNS by different routes, radiotherapy, IA carboplatin + radiotherapy was by far the best therapeutic modality in terms OS.

AIM - To conduct a phase I/II clinical study in which: (1) patients with relapsing GBM will be treated with a novel IA chemoradiation with Ca. (2) the new MRI sequence will be used to maximize the intraarterial catheter position in relation to individual tumor vasculature. Moreover, the investigators will assess whether the sequence can serve as a predictor of Ca delivery to the CNS, tumor response and patients survival. (3) Using tumor sample of each patient, to proceed to in vitro analysis of efflux pumps expression levels, DNA-bound Ca levels, and in vitro radiation linked to cell death study to predict in vivo tumor response. With this structuring and translational project, the investigators ultimate goal is to personalize GBM treatment for each patient based on the MRI and in vitro biological data.

HYPOTHESES - (1) IA Ca will show strong synergy with radiation and will act as a potent radiosensitizer. (2) MRI data analysis on blood flow, volume and vessel permeability will predict the extent of delivery of Ca to the tumor and the level of hypoxia affecting radiation effectiveness. Hence, this should allow to predict response to treatment. It will also help maximize the catheter position in the cerebral vascular tree. (3) In vitro intracellular penetration of carboplatin and radiation testing, as well as expression of efflux pumps will predict treatment effectiveness and time-correlate Ca binding to DNA with cell entrance flux. Putting together these data will allow correlating clinical and radiological response to quality of life (QOL), and to delivery surrogates for the IA infusion and intracellular penetration of carboplatin.

STUDY DESIGN: IA carboplatin and radiation - Patients with GBM progressing after the first line of treatment will be eligible. In this phase I/II trial, all patients will be treated at recurrence; a surgery will be performed for cytoreduction during which tumor samples will be collected, followed by a combination of radiation and IA Ca. A dose escalation protocol with consideration of the cumulative biologically effective dose and the normalized total dose will be used to determine the optimal re-irradiation dose in terms of acceptable toxicity and efficacy. We will use 10 fractions of radiation over 2 weeks. This will allow to benefit from the protective effects of fractionation (normal tissue repair), while being tolerable in the preservation of QOL. Escalation scheme from 1.5Gy/fraction up to 3.5Gy/fraction will allow to control for neurotoxicity. A 12 weeks observational period has been planned between each escalation to detect any undesired toxicity. Toxicity will be graded according to the National Cancer Institute (NCI) common toxicity criteria and grade III or IV will be considered significant. Pending the occurrence of such toxicity, the patient will be withdrawn from the study. Moreover, 3 instances of a grade III or IV toxicity will halt the escalation scheme. The prior radiation dose level will then be considered as the established safe level, and 10 more patients will be accrued at this level.

Combined with radiation, patients will receive 2 treatments of IA carboplatin12 (400 mg/m2), 4 hours prior to the first and the sixth radiation fraction (of a total of 10). IA treatments will then be continued on a monthly basis as a single treatment modality for consolidation, up to a total of 12 months, or until progression.

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of glioblastoma multiforme
2. Radiological progression on an MRI scan, according to the RANO criteria, in the context of a known glioblastoma multiforme, already treated with the Stupp protocol of combined radiotherapy-Temozolomide, and progressing. This implies a measurable disease on MRI.
3. Prior radiotherapy and temozolomide, as per the Stupp protocol, no sooner than 4 weeks, is permitted.
4. 18 of age and over
5. Performance status: Karnofsky 60-100%
6. Haematopoietic parameters at enrolment:

   * Platelet counts > 100,000/mm^3
   * Hemoglobin > 8 g/dL
   * Absolute neutrophil count > 1,500/mm^3
   * No impaired bone marrow function
7. Hepatic parameters at enrolment:

   * Bilirubin ≤ 2 times normal value
   * AST and ALT ≤ 2 times upper limit of normal (ULN) Alkaline phosphatase ≤ 2 times ULN (unless attributed to tumor)
   * No impaired hepatic function
8. Renal parameters at enrollment:

   * No impaired renal function
   * Creatinine no greater than 1.5 fold of the normal value
   * Creatinine clearance > 30 ml/min.
9. Normal ECG
10. Written informed consent obtained
11. Patient should be either sterile or else use a contraceptive strategy (for at least 2 months prior to study accrual).

    -

Exclusion Criteria:

1. Presence of a severe psychiatric or medical condition that would interfere with treatment administration or study enrolment.
2. Presence of an active auto-immune disease.
3. Occurrence of another malignancy within the past 5 years except curatively treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
4. Pregnancy (as objectivated by a positive b-HCG) or actively nursing
5. Presence of an uncontrolled systemic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2018-07-10 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
Response on MRI using the RANO Criteria | every 4 weeks until progression per RANO criteria
  T1, T2, FLAIR and a new diffusion protocol

SECONDARY OUTCOMES:
Incidence of treatment related Neurocognitive decline | Every 4 weeks until progression per RANO criteria
  MOCA questionnaire (Montreal Cognitive Assessment)
Quality of life (QOL) using SNAS questionnaire (Sherbrooke neuro assessment scale for quality of life). Scale range from 30 to 120; the lower scores indicate better quality of life. | Every 4 weeks until progression per RANO criteria
  SNAS Questionnaire
In vitro intracellular carboplatin accumulation | Once, 40 hours after surgery
  samples will then be analysed at one hour intervals for intracellular Pt concentration by Inductively Coupled Plasma Mass Spectrometer (ICP-MS). The amount of Pt bound to DNA will also be measured by ICP-MS. The level of apoptosis will be determined for each of the analysed sample

CONTACTS AND LOCATIONS:
Overall Officials: David Fortin, MD, Principal Investigator — CRC-CHUS
Locations (1):
- CHUS, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Charest G, Paquette B, Fortin D, Mathieu D, Sanche L. Concomitant treatment of F98 glioma cells with new liposomal platinum compounds and ionizing radiation. J Neurooncol. 2010 Apr;97(2):187-93. doi: 10.1007/s11060-009-0011-5. Epub 2009 Sep 17. PMID 19760366
- [Background] Goffaux P, Boudrias M, Mathieu D, Charpentier C, Veilleux N, Fortin D. Development of a concise QOL questionnaire for brain tumor patients. Can J Neurol Sci. 2009 May;36(3):340-8. doi: 10.1017/s0317167100007095. PMID 19534336
- [Background] Mathieu D, Fortin D. The role of chemotherapy in the treatment of malignant astrocytomas. Can J Neurol Sci. 2006 May;33(2):127-40. doi: 10.1017/s0317167100004881. PMID 16736721
- [Background] Charest G, Sanche L, Fortin D, Mathieu D, Paquette B. Glioblastoma treatment: bypassing the toxicity of platinum compounds by using liposomal formulation and increasing treatment efficiency with concomitant radiotherapy. Int J Radiat Oncol Biol Phys. 2012 Sep 1;84(1):244-9. doi: 10.1016/j.ijrobp.2011.10.054. Epub 2012 Jan 26. PMID 22284691
- [Background] Dea N, Fournier-Gosselin MP, Mathieu D, Goffaux P, Fortin D. Does extent of resection impact survival in patients bearing glioblastoma? Can J Neurol Sci. 2012 Sep;39(5):632-7. doi: 10.1017/s0317167100015377. PMID 22931705
- [Background] Daigle K, Fortin D, Mathieu D, Saint-Pierre AB, Pare FM, de la Sablonniere A, Goffaux P. Effects of surgical resection on the evolution of quality of life in newly diagnosed patients with glioblastoma: a report on 19 patients surviving to follow-up. Curr Med Res Opin. 2013 Oct;29(10):1307-13. doi: 10.1185/03007995.2013.823858. Epub 2013 Jul 30. PMID 23844725
- [Background] Charest G, Sanche L, Fortin D, Mathieu D, Paquette B. Optimization of the route of platinum drugs administration to optimize the concomitant treatment with radiotherapy for glioblastoma implanted in the Fischer rat brain. J Neurooncol. 2013 Dec;115(3):365-73. doi: 10.1007/s11060-013-1238-8. Epub 2013 Sep 13. PMID 24026531
- [Background] Drapeau A, Fortin D. Chemotherapy Delivery Strategies to the Central Nervous System: neither Optional nor Superfluous. Curr Cancer Drug Targets. 2015;15(9):752-68. doi: 10.2174/1568009615666150616123548. PMID 26077730
- [Background] Shi M, Fortin D, Sanche L, Paquette B. Convection-enhancement delivery of platinum-based drugs and Lipoplatin(TM) to optimize the concomitant effect with radiotherapy in F98 glioma rat model. Invest New Drugs. 2015 Jun;33(3):555-63. doi: 10.1007/s10637-015-0228-4. Epub 2015 Mar 18. PMID 25784204
- [Background] Fortin D, Morin PA, Belzile F, Mathieu D, Pare FM. Intra-arterial carboplatin as a salvage strategy in the treatment of recurrent glioblastoma multiforme. J Neurooncol. 2014 Sep;119(2):397-403. doi: 10.1007/s11060-014-1504-4. Epub 2014 Jun 20. PMID 24947313
- [Background] Blanchette M, Tremblay L, Lepage M, Fortin D. Impact of drug size on brain tumor and brain parenchyma delivery after a blood-brain barrier disruption. J Cereb Blood Flow Metab. 2014 May;34(5):820-6. doi: 10.1038/jcbfm.2014.14. Epub 2014 Feb 12. PMID 24517973